CLINICAL TRIAL: NCT04671160
Title: Impact of Continuous Veno-venous Hemodiafiltration on Efficacy of Administration of Prophylactic Doses of Enoxaparin or Fondaparinux in Critically Ill Patients.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Gdansk (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: M000000346978
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Assessment of Activity of Anti-Xa Factor in Patients Treated With Continuous Veno-venous Hemodiafiltration Receiving Anticoagulant Prophylaxis
Keywords: continuous veno-venous hemodiafiltration; enoxaparin; low molecular weight heparin; LMWH; CVVHDF; anticoagulant prophylaxis; critically ill; fondaparinux; anti-Xa activity
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: Group treated with CVVHDF and receiving enoxaparin as anticoagulant prophylaxis.
  Interventions: Diagnostic Test: Assessment the activity of anti-Xa factor.
- 2: Group treated with CVVHDF and receiving fondaparinux as anticoagulant prophylaxis.
  Interventions: Diagnostic Test: Assessment the activity of anti-Xa factor.
- 3: Group not treated with CVVHDF and receiving enoxaparin as anticoagulant prophylaxis.
  Interventions: Diagnostic Test: Assessment the activity of anti-Xa factor.
- 4: Group not treated with CVVHDF and receiving fondaparinux as anticoagulant prophylaxis.
  Interventions: Diagnostic Test: Assessment the activity of anti-Xa factor.

INTERVENTIONS:
Diagnostic Test: Assessment the activity of anti-Xa factor. — Assessment the activity of anti-Xa factor in patients treated with CVVHDF and receiving enoxaparin as anticoagulant prophylaxis, patients treated with CVVHDF and receiving fondaparinux as anticoagulant prophylaxis, patients not treated with CVVHDF and receiving enoxaparin as anticoagulant prophylaxis and patients not treated with CVVHDF and receiving fondaparinux as anticoagulant prophylaxis.

SUMMARY:
Dose of anticoagulant prophylaxis in patients with continuous veno-venous hemodiafiltration may be insufficient to keep anti-Xa factor activity in prophylactic range.

DETAILED DESCRIPTION:
Coagulation disorders are one of the most common complications in critically ill patients. Among them deep vein thrombosis and pulmonary embolism are the most significant factors increasing morbidity and mortality in ICU patients. Use of anticoagulant prophylaxis aims to prevent these dangerous complications. Most commonly used anticoagulant prophylaxis agents are low molecular weight heparins (LMWH). LMWH therapeutic efficiency is measured with activity of anti-Xa factor, that should range between 0.2 and 0.4 IU/mL in order to prevent thrombotic complications. Due to grave general condition, critically ill patients may often develop acute kidney injury (AKI), that requires renal replacement therapy (RRT). Because of haemodynamic instability the safest therapeutic choice seems to be continuous veno-venous hemodiafiltration (CVVHDF). This RRT mode removes particles in the size of few daltons even up to 10 kilodaltons (kDa) such as metabolic product waste, ions, hormones etc. LMWH with average molecular weight of 4.5 kDa and fondaparinux with average molecular weight of 1.7 kDa may be removed during CVVHDF resulting in insufficient activity of anti-Xa factor thus increasing the risk of thrombotic complications in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* All adult Intensive Care Unit patients between 18 and 80 years old requiring treatment with CVVHDF;
* Indications for anticoagulant prophylaxis with enoxaparin 40 mg sc. once daily or fondaparinux 2.5 mg sc. once daily;
* Treatment with continuous veno-venous hemodiafiltration.

Exclusion Criteria:

* Indications for low molecular weight heparin use other than anticoagulant prophylaxis;
* Intracranial hemorrhage;
* Incident of serious bleeding within a week before admission to ICU, if not managed;
* Disseminated intravascular coagulopathy;
* Heparin induced thrombocytopenia;
* Hypersensitivity or allergic reaction to enoxaparin or fondaparinux;
* Thrombocytopenia < 50 G/L;
* Prothrombin time < 20% or INR (international normalized ratio) > 1.7;
* Use of antiplatelet drugs;
* Presence of congenital coagulopathy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All male and female Intensive Care Unit adult patients (18 - 80 y.o.) requiring continuous veno-venous hemodiafiltration (CVVHDF) and receiving prophylactic doses of enoxaparin or fondaparinux.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-01-04 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Anti-Xa assay | 9 hours
  Anti-Xa assay as a tool to measure anticoagulation activity in subjects just before administration of anticoagulant prophylaxis, 3 hours, 6 hours and 9 hours after administration of prophylactic dose of enoxaparin 40 mg sc. once daily or fondaparinux 2.5 mg sc. once daily.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Gdansk - Departament of Anesthesiology and Intensive Care, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] Aszkielowicz A, Steckiewicz KP, Owczuk R. Evaluating the impact of continuous venovenous hemodiafiltration on the efficacy of prophylactic fondaparinux doses: a prospective single-center observational study. Sci Rep. 2025 May 24;15(1):18083. doi: 10.1038/s41598-025-03365-1. PMID 40413237